CLINICAL TRIAL: NCT00025389
Title: A Phase 2 Study Of Neoadjuvant rhuMAb VEGF (Bevacizumab) In Combination With Paclitaxel And Carboplatin In Surgically Resectable Non-Small Cell Lung Cancer
Brief Title: Bevacizumab, Paclitaxel, and Carboplatin Before Surgery in Treating Patients With Stage IB, Stage II, or Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12653A; UCCRC-12653A; NCI-2655; OSU-0120
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Bevacizumab (15mg/kg, q3wk x 2), Paclitaxel (200 mg/m2, q3wk x 2), carboplatin (AUC of 6, q3wk x 2), followed by surgery 4 to 6 weeks after last dose of Bevacizumab
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: paclitaxel
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy before surgery may may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is to see if bevacizumab, paclitaxel, and carboplatin given before surgery work in treating patients who have stage IB, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical complete and partial response rate in patients with stage IB, II, or IIIA resectable non-small cell lung cancer treated with neoadjuvant bevacizumab, paclitaxel, and carboplatin.
* Determine the pathologic complete response rate in patients treated with this regimen.
* Determine the ability to proceed with and complete a potentially curative resection in patients treated with this regimen.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: Patients receive neoadjuvant bevacizumab IV over 60-90 minutes, paclitaxel IV over 3 hours, and carboplatin IV over 1 hour on day 1.

Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgical resection within 4-6 weeks after completion of chemotherapy.

Patients are followed within 3 months.

PROJECTED ACCRUAL: A total of 23-39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IB (T2, N0), II (T1 or T2, N1 or T3, N0), or IIIA (T3, N1)
  * Potentially resectable disease
* No large central primary tumors in proximity to significant blood vessels
* No bronchoscopically evident endobronchial tumors
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy:

* More than 12 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of an inherited bleeding disorder
* No inherited predisposition to a hypercoagulable state
* No clinically evident hypercoagulable state or bleeding diathesis

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN
* INR less than 1.5
* PTT less than 36 seconds

Renal:

* Creatinine less than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min
* No nephrotic syndrome
* Urine protein no greater than 0.5 g/24 hours

Cardiovascular:

* No poorly controlled hypertension (greater than 150 mm Hg systolic and/or greater than 100 mm Hg diastolic) despite treatment
* No uncompensated coronary artery disease
* No myocardial infarction within the past 6 months
* No clinically significant or severe peripheral vascular disease
* No inherited predisposition to thrombosis
* No deep venous or arterial thrombosis
* No symptomatic congestive heart failure
* No unstable angina pectoris within the past 6 months
* No cardiac arrhythmia
* No transient ischemic attack within the past 6 months
* No cerebrovascular accident within the past 6 months
* No other arterial thromboembolic event within the past 6 months

Pulmonary:

* No hemoptysis
* No pulmonary embolism

Other:

* No history of allergic reactions to compounds of similar chemical or biologic composition to study drugs
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness or social situation that would preclude study compliance
* No significant traumatic injury within the past 28 days
* No uncontrolled concurrent illness
* No ongoing or active infection
* No serious, non-healing wound, ulcer, or bone fracture
* No other active malignancy
* No requirement for full-dose anticoagulation or thrombolytic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for this cancer
* No concurrent prophylactic growth factors (e.g., epoetin alfa, filgrastim [G-CSF], or sargramostim [GM-CSF])

Chemotherapy:

* No prior chemotherapy for this cancer
* Prior chemotherapy for another malignancy allowed provided the prior malignancy was curatively treated and is currently controlled

Endocrine therapy:

* No prior endocrine therapy for this cancer

Radiotherapy:

* No prior radiotherapy for this cancer
* Prior radiotherapy for another malignancy allowed provided the prior malignancy was curatively treated and is currently controlled
* No concurrent radiotherapy

Surgery:

* Prior diagnostic bronchoscopy, mediastinoscopy, or CT-guided biopsy allowed
* At least 28 days since prior major surgical procedure or open biopsy

Other:

* No other concurrent investigational agents
* No other concurrent anticancer investigational or commercial agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent low-dose warfarin for maintenence of preexisting, permanent, indwelling IV catheters allowed provided INR less than 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2001-11; Primary Completion 2005-12 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response Rate (complete and partial responses by RECIST) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Mauer, MD, Study Chair — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio